CLINICAL TRIAL: NCT06883552
Title: An Open-label, Single-arm Clinical Study of Stapokibart Injection in Combination with Tislelizumab Injection in Patients with Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM310_IIS_NSCLC08
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stapokibart Injection in Combination with Tislelizumab Injection in Patients with NSCLC (Experimental): During treatment cycles 1-18, Tislelizumab Injection will be administered in combination with Tislelizumab Injection. From cycle 19 onward, treatment will continue with Tislelizumab Injection monotherapy. The specific regimen is as follows:
  Tislelizumab Injection: 600 mg (initial dose) - 300 mg (subsequent doses), subcutaneously (SC), every 3 weeks (Q3W), for a total of 18 doses (1 year).
  Tislelizumab: 200 mg, intravenously (IV), every 3 weeks (Q3W).
  Interventions: Drug: Tislelizumab Injection

INTERVENTIONS:
Drug: Tislelizumab Injection — During treatment cycles 1-18, Tislelizumab Injection will be administered in combination with Tislelizumab Injection. From cycle 19 onward, treatment will continue with Tislelizumab Injection monotherapy. The specific regimen is as follows: Tislelizumab Injection: 600 mg (initial dose) - 300 mg (subsequent doses), subcutaneously (SC), every 3 weeks (Q3W), for a total of 18 doses (1 year). Tislelizumab: 200 mg, intravenously (IV), every 3 weeks (Q3W).

SUMMARY:
This is a single-arm study evaluating the efficacy and safety of Stapokibart Injection in combination with Tislelizumab Injection in patients with driver gene-negative NSCLC who have failed prior PD-1/PD-L1 inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Capable of comprehending the nature of the study and voluntarily signing the Informed Consent Form (ICF).
* Aged ≥18 and ≤75 years, regardless of gender.
* Patients with driver gene-negative NSCLC who have failed first-line standard therapy and are ineligible for second-line therapy or alternative chemotherapy regimens.
* Treatment failure definition: Disease progression during or after treatment. Changes in therapy due to drug intolerance are not considered treatment failure.
* At least one measurable tumor lesion per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Investigator-assessed life expectancy ≥3 months.
* Agreement to undergo tumor tissue biopsy prior to initial study treatment and during therapy when clinically feasible.
* Adequate organ function confirmed by laboratory tests within 7 days prior to first dose:

Bone marrow function (no transfusion/growth factors within 2 weeks pre-screening):

Absolute neutrophil count ≥1.5×10⁹/L;Platelet count ≥75×10⁹/L;Hemoglobin ≥90 g/L Hepatic function:Total bilirubin ≤1.5×ULN (≤3×ULN with liver metastases); AST/ALT ≤2.5×ULN (≤5×ULN with liver metastases);Albumin ≥28 g/L Renal function:Serum creatinine ≤1.5×ULN OR creatinine clearance ≥50 mL/min. Coagulation:INR and APTT ≤1.5×ULN. Chronic HBV-infected subjects must have HBV-DNA <1,000 IU/mL and commit to antiviral therapy throughout the study.

* Prior treatment-related toxicities resolved to ≤Grade 1 (CTCAE v5.0) or stabilized (excluding alopecia/pigmentation).
* Subjects of reproductive potential must use highly effective contraception from ICF signing until 6 months post-last dose.
* Ability to communicate effectively with investigators and comply with protocol-specified follow-up.

Exclusion Criteria:

* Received cytotoxic chemotherapy or Chinese herbal medicines with antitumor activity within 14 days prior to the first dose.
* Received radiotherapy, biologic therapy (e.g., cancer vaccines, cytokines, growth factors), or other immunotherapy (excluding PD-1/PD-L1 inhibitors) within 28 days or 5 half-lives (whichever is shorter) before the first dose.

Note: For palliative radiotherapy (≤14 days total duration) targeting non-CNS lesions, a ≥7-day washout period is required prior to the first dose.

* Received anti-interleukin-4 receptor alpha (IL-4Rα) monoclonal antibodies, anti-IgE monoclonal antibodies, or other biologics within 10 weeks or 5 half-lives (whichever is longer) before the first dose.
* Received live/attenuated vaccines within 12 weeks prior to the first dose or plans to receive such vaccines during the study.
* History of hypersensitivity to anti-IL-4Rα monoclonal antibodies, Stapokibart Injection, or other protein-based therapeutics (e.g., vaccines, immunoglobulins).
* Grade ≥3, severe, or life-threatening immune-related adverse events (irAEs) during prior immunotherapy (excluding Grade 3 endocrine AEs manageable with replacement therapy), or unresolved Grade 1-2 irAEs after treatment discontinuation.
* Clinically significant cardiovascular/cerebrovascular diseases, including:

Major events (e.g., congestive heart failure, acute MI, unstable angina, stroke, TIA, DVT/PE) within 6 months before the first dose.

* QTcF >480 msec.
* LVEF <50% by echocardiography.
* NYHA Class ≥2.
* Uncontrolled hypertension (SBP ≥160 mmHg or DBP ≥100 mmHg; rescreening permitted if controlled post-intervention).
* Other cardiovascular conditions deemed high-risk by investigators.
* Planned major surgery during the study period.
* Active CNS metastases. Note: Treated brain metastases may be eligible if radiographically/ clinically stable for ≥14 days before the first dose, confirmed by repeat imaging (≥4-week interval) during screening.
* Uncontrolled pleural, peritoneal, or pericardial effusion (investigator-assessed).
* Active Mycobacterium tuberculosis infection (i.e., active tuberculosis).
* HCV Ab-positive with detectable HCV RNA.
* HIV infection or positive HIV antibody test during screening.
* History of other malignancies within 5 years (exceptions: cured basal/squamous cell carcinoma, cervical/breast ductal carcinoma in situ).
* Active autoimmune disease requiring systemic treatment (e.g., immunomodulators, corticosteroids) within 2 years.

Note: Replacement therapy (e.g., thyroxine, insulin) is permitted.

* Prior organ or allogeneic hematopoietic stem cell transplantation.
* Pregnancy or lactation.
* Any condition that may confound study results, impair compliance, or jeopardize subject safety (investigator-determined).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to approximately 2 years
  Proportion of subjects with the best overall response (BOR)

SECONDARY OUTCOMES:
DOR | Up to approximately 2 years
  DOR is the time between the first observed tumor responseto disease progression or relapse based on RECIST Version 1.1
DCR | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1
PFS | Up to approximately 2 years
  PFS is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
OS | Up to approximately 2 years
  OS is the time from the date of randomization or first dosing date to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Wang, Principal Investigator — West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes